CLINICAL TRIAL: NCT02593565
Title: The Vasculitis Pregnancy Registry (V-PREG)
Brief Title: Vasculitis Pregnancy Registry
Acronym: V-PREG
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Duke University (Other); University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: VCRC 5532
Record Dates: First submitted 2015-10-26; First posted 2015-11-02 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Vasculitis; Behcet's Disease; CNS Vasculitis; Cryoglobulinemic Vasculitis; Eosinophilic Granulomatosis With Polyangiitis (EGPA); Churg-Strauss Syndrome (CSS); Granulomatosis With Polyangiitis (GPA); Wegener's Granulomatosis; IgA Vasculitis; Henoch-Schoenlein Purpura (HSP); Microscopic Polyangiitis (MPA); Polyarteritis Nodosa (PAN); Takayasu Arteritis (TAK); Urticarial Vasculitis; Systemic Vasculitis
MeSH Terms: conditions — Vasculitis; Behcet Syndrome; Vasculitis, Central Nervous System; Cryoglobulinemia, Familial Mixed; Churg-Strauss Syndrome; Granulomatosis with Polyangiitis; IgA Vasculitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis; Systemic Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intervention: Woman, 18 years of age or older, currently pregnant, and have a diagnosis of vasculitis.
  Interventions: Other: Online questionnaires

INTERVENTIONS:
Other: Online questionnaires — Women will be asked to complete questionnaires during their pregnancy and a postpartum questionnaire.

SUMMARY:
The purpose of this study is to learn about the experience of women with vasculitis who become pregnant. In particular, the study will consist of several online surveys to assess

1. each woman's vasculitis severity and pregnancy-related experiences, and
2. pregnancy outcomes.

DETAILED DESCRIPTION:
The study will consist of several on-line surveys to assess each woman's vasculitis severity, pregnancy-related experiences, and pregnancy outcomes. Participants will be asked to complete questionnaires at study entry, during the second trimester, during the third trimester, and postpartum. Investigators estimate that it will take approximately 20 minutes to complete each survey. The survey is available in Spanish, Portuguese, Italian, and Turkish.

All women enrolled in the Vasculitis Patient-Powered Research Network (VPPRN) (with specified disease, sex, and age inclusion criteria described below) will be invited via email to participate in this on-line study. The survey data will be stored by the Data Management and Coordinating Center (DMCC) at the University of South Florida. Upon conclusion of the study period, the data will be sent to the Study Chairs.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years of age or older with one of the following diseases may take part in the study:

   * Behçet's disease;
   * Central nervous system (CNS) vasculitis;
   * Cryoglobulinemic vasculitis (Cryoglobulinemia);
   * Eosinophilic granulomatosis with polyangiitis (also called Churg-Strauss Syndrome);
   * Giant Cell (Temporal) Arteritis (GCA);
   * Granulomatosis with polyangiitis (also called Wegener's);
   * IgA vasculitis (Henoch-Schoenlein purpura);
   * Microscopic polyangiitis (MPA);
   * Polyarteritis nodosa (PAN);
   * Takayasu's arteritis (TAK);
   * Urticarial vasculitis;
   * Other/Suspected Diagnosis.
2. Women must be pregnant (self-report) at the time of enrollment into the registry.

Exclusion Criteria:

1. Non-English speaking, with the exception of people who speak Spanish, Portuguese, Italian, or Turkish.
2. Unable to provide consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with vasculitis who are currently pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Unique pregnancy characteristics among women with vasculitis. | Four years
  To understand pregnancy characteristics and outcomes among women with vasculitis using patient-reported questionnaires in each trimester.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Clowse, MD, MPH, Study Chair — Duke University; Peter A Merkel, MD, MPH, Study Chair — University of Pennsylvania
Locations (1):
- University of South Florida Data Management and Coordinating Center, Tampa, Florida, United States

REFERENCES:
- [Result] Sims CA, Eudy AM, Larson K, Yeung C, Tam H, Kullman J, Borchin RL, Burroughs C, Merkel PA, Clowse MEB; VPREG Collaborative Group. Reproductive Outcomes for Women With Vasculitis. J Rheumatol. 2024 Oct 1;51(10):1003-1008. doi: 10.3899/jrheum.2023-1246. PMID 38825354
- [Result] Sims CA, Perry B, Yeung C, Tam H, Kullman J, Borchin RL, Burroughs C, Merkel PA, Clowse MEB. Exploring Reproductive Experiences With Women Enrolled in the International Vasculitis Pregnancy Registry. J Rheumatol. 2024 Oct 1;51(10):997-1002. doi: 10.3899/jrheum.2023-1055. PMID 38825350
- See also: The Vasculitis Patient-Powered Research Network — http://vpprn.org
- See also: Vasculitis Pregnancy Registry (VPREG) Information — https://www.vasculitisfoundation.org/vpreg/